CLINICAL TRIAL: NCT02571829
Title: A Phase II Single Arm Study Assessing Efficacy & Safety of Ribociclib in Patients With Advanced Well-Differentiated or Dedifferentiated Liposarcoma
Brief Title: A Phase II Study Assessing Efficacy & Safety of Ribociclib in Patients With Advanced Well/Dedifferentiated Liposarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Daniela Katz, MD, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEE011-HMO-CTIL
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Liposarcoma; Soft Tissue Sarcoma
Keywords: Liposarcoma; Soft tissue sarcoma; CDK4; CDK6; LEE011; ribociclib
MeSH Terms: conditions — Liposarcoma; Sarcoma | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ribociclib (Experimental): single arm ribociclib Oral 600 mg x 1 a day duration according to response.
  Interventions: Drug: ribociclib

INTERVENTIONS:
Drug: ribociclib — Oral, 600 mg x 1 a day, duration - according to response
  Other Names: LEE011

SUMMARY:
The purpose of this study is to determine whether ribociclib are effective and safe in the treatment of progressive well/dedifferentiated liposarcoma (WDL/DDL).

DETAILED DESCRIPTION:
The expected duration of this study is 36 months (24 months accrual period and 12 month follow up period). Enrollment into the screening or treatment phase of the study will be stopped when the actual subject numbers have been achieved.

This single arm single institution, open label, prospective, phase II trial will evaluate the efficacy and safety of oral 600mg/daily in 28 day cycles of ribociclib in advanced well-differentiated liposarcoma (WDL) and de-differentiated liposarcoma (DDL) patients. Number of patients in the study will reflect the reconciliation between statistical requirements and incidence.

Treatment will continue until disease progression, development of unacceptable toxicity, noncompliance or withdrawal of consent by the patient or investigator decision.

All screening requirements must be completed within 28 days of the visit (except for CDK4/6 amplification and pRb, p16 and cyclin D staining status which may be completed in advance). Patients will be examined on cycle 1 day-1 and every 2 weeks, including complete blood count (CBC) and chemistry, for the first 8 weeks of treatment, and thereafter every month until disease progression. CT/MRI imaging (contrast) will be performed every 8 weeks for response evaluation. Clinical benefit as well as individual categories of response (complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD) will be determined using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST). Response duration endpoints, including PFS, PFS at 12 weeks and OS will be assessed using the Kaplan-Meier method. Toxicity (AEs) will be recorded using the NCI- Common Toxicity Criteria for Adverse Effects v 4.03 (NCI-CTCAE). Screening procedures will include quantitative analysis of CDK4 gene copy number using FISH, immunostaining for p16 and cyclin D1 all using formalin fixed paraffin embedded (FFPE) tissue sections. In addition tumor DNA, extracted from FFPE tissue (after choosing optimal area by a Pathologist), will be submitted to a next generation sequencing analysis ("ion ampliseq" cancer panel v2©) for a later exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age ≥ 18 years
3. Histological confirmed diagnosis of WDL/DDL with metastatic or locally advanced disease not amenable to complete resection.
4. WDL/DDL patients must have documentation of disease progression within 6 months prior to study entry.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. Measurable disease by RECIST v1.1 criteria. At least one measurable lesion located outside of a previously irradiated area.
7. Formalin fixed paraffin embedded tumor blocs and representative hematoxylin/eosin slides (preferably both) should be provided for immunohistochemistry staining and molecular analysis of 50 gene signature panel and must have increased CDK4 gene copy number (at least >/=3) and proficient Rb gene.
8. Patient has adequate bone marrow and organ function.
9. Must be able to swallow ribociclib capsules/tablets.

Exclusion Criteria:

1. A known hypersensitivity to ribociclib or any of its excipients.
2. A concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
3. Patients with central nervous system (CNS) involvement at least 4 weeks from prior therapy completion
4. Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality within 12 months of screening)
5. On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF >450 msec
6. Participation in a prior investigational study within 30 days prior to enrollment
7. Patient has had major surgery within 14 days prior to starting study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Response to therapy as evaluated by RECIST 1.1 and Choi | 36 months (24 months accrual period and 12 month follow up period)

SECONDARY OUTCOMES:
Median PFS and PFS assessed at 12 weeks (PFS will be computed from the date of start of treatment to the first documented date of progression or the date of death, due to any cause assessed by investigator. | 12 weeks
Overall survival (OS) will be computed from the date of start of treatment to the date of death, due to any cause. Patients alive or lost for follow-up at the time of the analysis will be censored at the date of last follow-up. | 36 months (24 months accrual period and 12 month follow up period)
Evaluate the time from first documented response to disease progression | 36 months (24 months accrual period and 12 month follow up period)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Katz, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Shapiro GI. Cyclin-dependent kinase pathways as targets for cancer treatment. J Clin Oncol. 2006 Apr 10;24(11):1770-83. doi: 10.1200/JCO.2005.03.7689. PMID 16603719
- [Background] Ortega S, Malumbres M, Barbacid M. Cyclin D-dependent kinases, INK4 inhibitors and cancer. Biochim Biophys Acta. 2002 Mar 14;1602(1):73-87. doi: 10.1016/s0304-419x(02)00037-9. PMID 11960696
- [Background] Barretina J, Taylor BS, Banerji S, Ramos AH, Lagos-Quintana M, Decarolis PL, Shah K, Socci ND, Weir BA, Ho A, Chiang DY, Reva B, Mermel CH, Getz G, Antipin Y, Beroukhim R, Major JE, Hatton C, Nicoletti R, Hanna M, Sharpe T, Fennell TJ, Cibulskis K, Onofrio RC, Saito T, Shukla N, Lau C, Nelander S, Silver SJ, Sougnez C, Viale A, Winckler W, Maki RG, Garraway LA, Lash A, Greulich H, Root DE, Sellers WR, Schwartz GK, Antonescu CR, Lander ES, Varmus HE, Ladanyi M, Sander C, Meyerson M, Singer S. Subtype-specific genomic alterations define new targets for soft-tissue sarcoma therapy. Nat Genet. 2010 Aug;42(8):715-21. doi: 10.1038/ng.619. Epub 2010 Jul 4. PMID 20601955
- [Background] Dickson MA, Tap WD, Keohan ML, D'Angelo SP, Gounder MM, Antonescu CR, Landa J, Qin LX, Rathbone DD, Condy MM, Ustoyev Y, Crago AM, Singer S, Schwartz GK. Phase II trial of the CDK4 inhibitor PD0332991 in patients with advanced CDK4-amplified well-differentiated or dedifferentiated liposarcoma. J Clin Oncol. 2013 Jun 1;31(16):2024-8. doi: 10.1200/JCO.2012.46.5476. Epub 2013 Apr 8. PMID 23569312
- [Background] Van Glabbeke M, Verweij J, Judson I, Nielsen OS; EORTC Soft Tissue and Bone Sarcoma Group. Progression-free rate as the principal end-point for phase II trials in soft-tissue sarcomas. Eur J Cancer. 2002 Mar;38(4):543-9. doi: 10.1016/s0959-8049(01)00398-7. PMID 11872347